CLINICAL TRIAL: NCT06263088
Title: EQUITY GI: A Prospective Study to Enhance Quality, Inclusivity, and Trial Participation in Black Patients With Gastrointestinal Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE15223
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Cancer; Colon Cancer; Rectal Cancer; Anal Cancer; Esophageal Cancer; Stomach Cancer; Appendix Cancer; Pancreas Cancer; Liver Cancer; Neuroendocrine Tumors
Keywords: Gastrointestinal cancer; African Americans
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Appendiceal Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Single arm study to address the existing disparities faced by Black participants with gastrointestinal (GI) cancer in accessing crucial biomarker testing, receiving evidence-based care, and participating in clinical trials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EQUITY GI (Other): 1. Data gathering
  2. Program development and implementation
  3. Health literacy
  Interventions: Other: EQUITY GI

INTERVENTIONS:
Other: EQUITY GI — 1. Ensuring appropriate biomarker testing and evidence-based care: Biomarker testing can also help choose treatment. Additionally, a tumor board will be conducted periodically to provide treatment recommendations to the treating physician. Participant will receive standard-of-care treatment if they enroll in this study. Participant will not receive any experimental treatment.
  2. Assistance with clinical trial enrollment. The study team will help enroll in a clinical trial appropriate for the condition.
  3. Health literacy: The study team will provide information relevant to your diagnosis to enrich your understanding of your condition and treatment. Investigator will provide questionnaires to assess your understanding before and after you have been provided with educational/informational material appropriate for your diagnosis.

SUMMARY:
This research study is being conducted to improve the quality of care of participants who have a diagnosis of gastrointestinal cancer (anal, colon, rectal, esophageal, stomach, small bowel, appendix, pancreas, gall bladder, liver, neuroendocrine tumor of gastrointestinal origin).

This study has 3 components as follows-

1. Ensuring appropriate biomarker testing and evidence-based care: Biomarkers are molecules in the tumor or blood that indicate normal or abnormal processes in participant's body and may indicate an underlying condition or disease. Various molecules, such as DNA (genes), proteins, or hormones, can serve as biomarkers since they all indicate something about participant's health. Biomarker testing can also help choose participant's treatment. Additionally, a tumor board will be conducted periodically to provide treatment recommendations to participant's treating physician. Participants will receive standard-of-care treatment if participant enroll in this study. Participant will not receive any experimental treatment.
2. Assistance with clinical trial enrollment. The study team will help participants enroll in a clinical trial appropriate for participant's condition. However, enrolling in a clinical trial is totally up to the participant.
3. Health literacy: The study team will provide information relevant to participant's diagnosis to enrich participant's understanding of participant's condition and treatment. Investigator will provide questionnaires to assess participant's understanding before and after participant's have been provided with educational/informational material appropriate for participant's diagnosis.

DETAILED DESCRIPTION:
Black individuals, including African Americans, have a disproportionate cancer burden, including the highest mortality and the lowest survival of any racial/ethnic group for most cancers.1 Colorectal cancer (CRC), the most common subtype of GI cancer, is the third most frequently diagnosed cancer among Black men and women.1 Black participants have a disproportionate gastrointestinal (GI) tract cancer burden compared with White participants, with a 19% excess risk of cancer death for men and a 13% excess risk for women.2 Almost two decades after the Institute of Medicine's Unequal Treatment report,3 the treatment gap persists among Black participants with GI cancer across treatment settings and modalities.4 A National Cancer Database (NCDB)-based analysis suggests that Black participants with GI cancers are less likely than White participants to achieve negative surgical margins, undergo adequate lymphadenectomies, and less often receive adjuvant therapies.4 Similar data demonstrates racial disparities in care and outcomes in many GI cancer types.5-8 It is important to emphasize that the disparity of cancer care among Black participants shown in the published studies is likely an underestimate given that Black participants are less likely to receive appropriate workups leading to a cancer diagnosis because of the mistrust in the existing system.9 The age-standardized incidence of various GI cancers, including colon, rectal, liver, intrahepatic bile duct, stomach, and pancreatic cancers, is projected to rise in the United States (US) in the coming decades,10 strongly supporting a need for innovative measures to address the care gap. With this proposed project, investigator seeks to address this troubling disparity by assessing the extent of the care gap, expanding the biomarker testing and evidence-based care through the molecular tumor board, and implementing a information platform integrated with EPIC electronic health record system that will guide providers to navigate the biomarker-driven therapy and clinical trial enrollment.

University Hospitals Seidman Cancer Center (UH SCC) is a large hybrid academic-community oncology network that includes the main academic center and 15 community-based cancer centers. At UH SCC, approximately 2000 participants with GI cancer diagnoses are treated annually, and 15 % of these participants are Black. Investigator retrospectively reviewed all cases of CRC, the most prevalent GI cancer, diagnosed in the UH SCC system from April 2020 to March 2022 and found that only 30% of participants underwent all appropriate biomarker testing. Biomarker testing rates were particularly low in community sites. In addition, approximately 15% of participants treated for CRC at UH SCC were underserved minorities, predominantly Black, in whom the rate of biomarker testing was even lower (20%). These data highlight the urgent need for measures to close the care gap. Our colleagues at UH SCC in the thoracic oncology group previously demonstrated the feasibility of improving biomarker testing and implementing biomarker-guided treatment by utilizing an integrated information platform that tracks the biomarker test results.11 Investigator plans to create a similar integrated information platform for GI cancer participants, 'EQUITY GI Oncotracker.'

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old.
2. Newly diagnosed Black GI cancer participants irrespective of stage. Eligible tumor types include anal carcinoma, rectal cancer, colon cancer, small bowel cancer, appendix carcinoma, hepatobiliary cancer, pancreatic cancer, gastroesophageal cancer, gastrointestinal neuroendocrine tumors, and gastrointestinal stromal tumor.
3. Patient able and willing to comply with study procedures
4. The patient is able to understand and willing to sign and date the written informed consent form at the screening visit.

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker testing rate of Black participants diagnosed with GI cancer | 24 months
  The biomarker testing rate will be estimated based on the number of cases (i.e., participants taking the biomarker testing) using a binomial distribution, and their confidence intervals will be estimated using Wilson's method.23 Potential predictors of the binary outcomes will be identified using multivariable logistic regression.

SECONDARY OUTCOMES:
Clinical trial enrollment rate among black participants diagnosed with GI cancer | 24 months
  The clinical trial enrollment rate will be estimated based on the number of cases (i.e., participants enrolled in clinical trials) using a binomial distribution, and their confidence intervals will be estimated using Wilson's method.23 Potential predictors of the binary outcomes will be identified using multivariable logistic regression.
Change in Health literacy test among black participants diagnosed with GI cancer | 24 months
  The evaluation of literacy will be conducted using the CHLT-6 questionnaire, a six-item test designed for assessing cancer health literacy measured before and after the intervention with the goal of increasing the mean score by 30%.
Change in Health literacy score among black participants diagnosed with GI cancer | 24 months
  The evaluation of literacy will be conducted using the CHLT-30 questionnaire, a thirty-item test designed for assessing cancer health literacy measured before and after the intervention with the goal of increasing the mean score by 30%.

CONTACTS AND LOCATIONS:
Overall Officials: Sakti Chakrabarti, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Until 2026